CLINICAL TRIAL: NCT01186835
Title: Treatment of Forehead/Glabellar Rhytide Complex With Combination Botulinum Toxin A and Hyaluronic Acid Versus Botulinum Toxin A Injection Alone: A Split-face, Rater-blinded Randomized Control Trial
Brief Title: Treatment of Forehead/Glabellar Rhytide Complex With Combination Botulinum Toxin A and Hyaluronic Acid Versus Botulinum Toxin A Injection Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Principal Investigator, Murad Alam, Associate Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MA-stu24810
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Forehead/Glabellar Rhytid Complexes
MeSH Terms: interventions — Hyaluronic Acid; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Botulinum Toxin A and Hyaluronic Acid (Experimental): One side of face treated with the combination of Botulinum Toxin A and Hyaluronic Acid injections.
  Interventions: Procedure: Combination Botulinum Toxin A and Hyaluronic Acid
- Botulinum Toxin A alone (Active Comparator): Other side of face treated with =Botulinum Toxin A injection alone.
  Interventions: Procedure: Botulinum Toxin A

INTERVENTIONS:
Procedure: Combination Botulinum Toxin A and Hyaluronic Acid — One side of subject's face will randomly be assigned combination treatment.
  Arms: Combination Botulinum Toxin A and Hyaluronic Acid
Procedure: Botulinum Toxin A — Other side of subjects face with receive Botulinum Toxin A treatment alone.
  Arms: Botulinum Toxin A alone

SUMMARY:
The objective of this study is to determine whether the use of botulinum toxin (Dysport ®) in conjunction with a hyaluronic acid filler (Restylane®) will improve the appearance of wrinkles on the forehead and glabella (area between the eyebrows) better than botulinum toxin alone. These two products have been FDA approved to improve the appearance of facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Is 18-65 years of age
* Has static and dynamic forehead/glabellar wrinkles
* Has willingness and the ability to understand and provide informed consent and communicate with the investigator

Exclusion Criteria:

* Pregnant or lactating
* Has received the following treatments in the forehead or glabellar region:

  * botulinum toxin injections in the past 6 months
  * ablative laser procedure in the past 6 months
  * radiofrequency device treatment in the past 6 months
  * ultrasound device treatment in the past 6 months
  * medium to deep chemical peel in the past 6 months
  * temporary soft tissue augmentation material in the past year
  * semi-permanent soft tissue augmentation material in the past 2 years
  * permanent soft tissue augmentation material
* Is planning to receive within the next 6 months, any cosmetic procedure (such as any chemical peels, botulinum toxin injections, ablative or non-ablative laser procedures, filler injections, radiofrequency procedures, dermabrasion, ultrasound and face lifting procedures) in the forehead or glabellar region.
* Is planning to use tretinoin or retinoic acid in the next 6 months
* Has an active infection in the forehead or glabellar region (excluding mild acne)
* Is allergic to cow's-milk protein
* Is allergic to albumin
* Taking aminoglycoside
* Has prior history of nodule formation or hypersensitivity reactions to lidocaine or hyaluronic acid derivatives
* Is currently using anticoagulation therapy
* Has a history of bleeding disorders
* Is unable to understand the protocol or to give informed consent
* Has a mental illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Measure: | 1 year
  Two blinded dermatologists will rate each photograph of each subject at baseline, week 2, month 3, and month 6. The raters will provide a glabellar wrinkle score and a forehead wrinkle score for each photograph. The raters will not know what treatments the subjects received or at what point in time the photographs were taken.

SECONDARY OUTCOMES:
Measure: Percent Improvement | 1 year
  * Two blinded dermatologists will also rate the percent improvement between the before and after photographs (Appendix III).
  * A live blinded dermatologist will determine which side looks better at week 0, week 2, month 3, and month 6.
  * A subject self-evaluation will be administered at week 2, month 3, and month 6.
  * A subject satisfaction questionnaire will be administered at month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Alejandra Onate, Chicago, Illinois, United States